CLINICAL TRIAL: NCT04633083
Title: Range of Motion Analysis for the Optimization of Reverse Shoulder Arthroplasty Planning
Brief Title: Range-of-motion Analysis of Reverse Shoulder Arthroplasty
Acronym: ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S62153
Record Dates: First submitted 2019-01-22; First posted 2020-11-18 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Signs of impingement (Other): a. non- limited ROM i. Endorotation control until lumbosacral level ii. Scapular plane abduction above 150° b. limited ROM i. Endorotation control lower then lumbosacral level ii. Scapular plane abduction under 150°
  Intervention: clinical data, imaging data, movement analysis, EOS measurements, ROM simulation
  Interventions: Other: Data collection
- No Signs of impingement (Other): a. non- limited ROM i. Endorotation control until lumbar level ii. Scapular plane abduction above 150° b. limited ROM i. Endorotation control lower then lumbar level ii. Scapular plane abduction under 150°
  Intervention: clinical data, imaging data, movement analysis, EOS measurements, ROM simulation
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Clinical Data: Registration of patient identity, sex and birth year, Body Mass Index, generic score EQ-5D-3L, Tampa Schaal voor kinesofobia and shoulder specific score like Constant Score, PROMS, ADLER, SST and postoperative ROM.
  Imaging Data: A preoperative and postoperative CT scan and 1-year postoperative radiograph (all three part of standard clinical practice) will be obtained. This data is used to extract the bone geometries and implant position.
  Movement Analysis: The subject should stand still followed by different motion tasks in the gait lab with collection of shoulder girdle kinematics and kinetics using a 14-camera VICON System.
  Stereo Radiographic EOS Measurements: Every subject included in the study will undergo a stereo radiographic EOS exam while quite standing with their arm in various positions (van Andel et al., 2008) .
  ROM simulation: With the developed ROM software, we will simulate the ROM of the 2 patient groups based on the available CT scan data.

SUMMARY:
Limited range-of-motion (ROM) is a common problem after reverse shoulder arthroplasty (RSA). The occurrence and magnitude depend on both surgical and patient-related factors. The most important surgical factor is the occurrence of impingement, which implicates collision between the humeral implant or bone and the scapula, limiting further motion. Patient-related factors such as scapula geometry and muscle function and activation also play an important role. Surgeons have to account for these factors when planning and implanting a RSA. Software models can support the surgeon during preoperative planning by using imaging data to simulate the ROM of a patient's shoulder after RSA. These software models allow for adaptation of the implant position during preoperative planning and, by this optimize the postoperative ROM. However, the models currently developed are limited in terms of ROM simulation and the factors the models take into account.

DETAILED DESCRIPTION:
The impingement-free ROM in a RSA patient is defined as the rotational area the humeral liner can move through without colliding against the scapula or dislocating the joint. In a previous study, a new software model was developed that uses imaging data to compute and quantify the impingement-free ROM of a patient according to clinically relevant motions. Before this model can be used in clinical practice, a validation of the model's accuracy in predicting real RSA patient outcomes is required. Therefore, the first objective is to verify the model's ability to predict the ROM of the glenohumeral joint in real RSA patients. The investigators will investigate and quantify the ROM and joint angles of RSA patients with and without impingement with the help of EOS imaging and video motion analysis. The investigators can then compare model outputs with measured patient outcomes. Additionally, the investigators will investigate how well our software model can predict impingement in patients with known postoperative impingement.

Currently, the software model uses a database of healthy shoulder kinematic motions to produce an objective ROM score for a RSA. However, it is not known if healthy shoulder kinematics are a suitable reference for quantifying and interpreting RSA kinematics. Glenohumeral motions of healthy subjects are already extensively described by Ludewig et al. Glenohumeral motions of RSA patients are not yet reported. Also, little is known about muscle activation patterns in RSA patients. The second objective is to describe muscle activation patterns and shoulder kinematics of RSA patients and compare our measured RSA kinematic motions to the healthy kinematic motion data currently used in the software model. Therefore, the investigators will perform instrumented 3D motion analysis in conjunction with electromyography measurements to incorporate muscle activation patterns into our RSA glenohumeral motion analysis. Our additional sub-objective is to compare muscle activation patterns between patients with and without limited ROM, with the goal of identifying differences between the two groups.

The third objective is to identify patient-related and implant related factors that influence the ROM after a reversed shoulder arthroplasty. Therefore, the investigators will investigate clinical factors that could have effect on the ROM after RSA. The different factors (sex, birth year, Body Mass Index, generic score EQ-5D-3L, Tampa Schaal voor kinesofobia) will be analyzed both across and within patients with and without limited ROM with the goal of identifying their relation to ROM. The most important implanted related factor will also be investigated and analyzed both across and within groups: implant position in terms of glenoid component version, inclination and location of center of rotation.

ELIGIBILITY:
Inclusion Criteria:

* Adults with RSA operated in the University Hospitals Leuven, Belgium
* Ability and willingness of patient to attend follow-up visit and complete patient questionnaires
* Complete patient informed consent
* Preoperative CT-scan available
* Pain free RSA (VAS score ≤ 3) more than 1 year postoperative

Exclusion Criteria:

* Only RSA patients with a functional RSA will be included, so patients with postoperative stiffness, pain, instability or pseudoparalysis will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Demographic data (Sex) | 1-time assessment at a time of 1 or more years postoperatively
  Sex
Demographic data (Birth year) | 1-time assessment at a time of 1 or more years postoperatively
  Birth year
Demographic data (Body Mass Index) | 1-time assessment at a time of 1 or more years postoperatively
  Body Mass Index in kg/m2 (physiological parameter)
Demographic data (Range of motion) | 1-time assessment at a time of 1 or more years postoperatively
  Range of motion in degrees (physiological parameter)
Imaging data | 1-time assessment at a time of 1 or more years postoperatively
  Pre- and post-surgery CT scan
Movement analysis | 1-time assessment at a time of 1 or more years postoperatively
  The subject should stand still followed by different motion tasks in the gait lab with collection of shoulder girdle kinematics and kinetics using a 14-camera VICON System
Stereo Radiographic EOS Measurements | 1-time assessment at a time of 1 or more years postoperatively
  Every subject included in the study will undergo a stereo radiographic EOS exam while quite standing with their arm in various positions (van Andel et al., 2008)
ROM simulation | 1-time assessment at a time of 1 or more years postoperatively
  Simulate the ROM of the 2 patient groups based on the available CT scan data
EQ-5D-3L questionnaire | 1-time assessment at a time of 1 or more years postoperatively
  It is a questionnaire to measure health-related quality of life
Tampa scale for kinesiophobia (fear of movement) | 1-time assessment at a time of 1 or more years postoperatively
  It is a questionnaire that gives an impression of the degree of pain-related fear in patients with low back pain (LBP) or fibromyalgia.
Constant Score | 1-time assessment at a time of 1 or more years postoperatively
  These parameters define the level of pain and the ability to carry out the normal daily activities of the patient
ADLER (Activities of Daily Living [ADL] which require active External Rotation [ER]) | 1-time assessment at a time of 1 or more years postoperatively
  It measures the severity of the potential handicap
SST (Simple Shoulder Test) | 1-time assessment at a time of 1 or more years postoperatively
  It is a measuring instrument that measures the functional limitations of the affected shoulder of patients with shoulder complaints

CONTACTS AND LOCATIONS:
Overall Officials: Filip Verhaegen, MD, Principal Investigator — Medical Doctor, Principal Investigator
Locations (1):
- UZ Leuven, campus Pellenberg, Pellenberg, Belgium

IPD SHARING:
Plan to Share IPD: No